CLINICAL TRIAL: NCT06517966
Title: RUDRA Registry (Real-World Clinical Registry for Patients With Recurrent Pericarditis)
Status: Active, not recruiting | Type: Observational
Sponsor: Eurasian Association of Therapists (Other)
Responsible Party: Sponsor
Other Study IDs: RUDRA
Record Dates: First submitted 2024-07-15; First posted 2024-07-24 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Pericarditis
MeSH Terms: conditions — Pericarditis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Retrospective branch: All patients diagnosed with recurrent pericarditis within the previous 10 years (of any genesis) were included.
- Prospective branch: All patients with one of the following conditions were included:
  * a specialist-confirmed diagnosis of "recurrent pericarditis" without an established etiology at the time of inclusion in the study (suspected "idiopathic recurrent pericarditis");
  * a specialist-confirmed diagnosis of idiopathic recurrent pericarditis.

SUMMARY:
А multicenter, non-interventional real world clinical registry of patients with recurrent pericarditis.

The main goal of the registry is to epidemiologically assess the pattern, clinical outcomes, and approaches to therapy in patients with recurrent pericarditis.

DETAILED DESCRIPTION:
А multicenter, non-interventional real world clinical registry of patients with recurrent pericarditis.

The main goal of the registry is to epidemiologically assess the pattern, clinical outcomes, and approaches to therapy in patients with recurrent pericarditis.

This goal can best be achieved through a registry of real clinical practice. Epidemiologic assessment of the structure will be possible due to the retrospective part of the registry and will give an idea of the etiology of RP in the Russian Federation, as well as allow to identify a subpopulation of patients with idiopathic recurrent pericarditis and study it in more detail. The prospective branch involves three-year dynamic follow-up of patients with already diagnosed and newly diagnosed IRP. Based on the data obtained during the retro- and prospective parts of the registry, it will be possible to evaluate clinical outcomes and approaches to therapy in patients with recurrent pericarditis, which may become valuable material for assessing the real clinical situation in the Russian Federation, as well as deepen knowledge on the diagnosis and management of this cohort of patients.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women 18 years of age or older at the time of data recording or pericarditis debut;
2. Presence of one of the following conditions:

   * a specialist-confirmed diagnosis of recurrent pericarditis without an established etiology at the time of inclusion in the study (suspected "idiopathic recurrent pericarditis");
   * a specialist-confirmed diagnosis of "idiopathic recurrent pericarditis".

Exclusion Criteria:

1. Age below 18 years at the time of inclusion in the registry or debut of pericarditis;
2. Specialist-confirmed secondary genesis of RP (infectious, autoimmune, neoplastic, metabolic, traumatic, iatrogenic, etc.); 2. Manifestations and complications of myocarditis, various diseases of thoracic organs, systemic diseases, cardiac surgery, radiation therapy, tuberculosis, etc.);
3. lack of possibility of screening examination and dynamic follow-up;
4. Organ/tissue transplantation less than 5 years prior to study inclusion or debut of pericarditis;
5. Oncologic disease less than 3 years prior to study inclusion or pericarditis debut;
6. Chemotherapy with anthracycline-type drugs at the time of pericarditis debut;
7. Administration of amphetamine-type drugs at the time of pericarditis debut;
8. Cardiac/pericardial surgery in the last 6 months prior to study inclusion or pericarditis debut;
9. Myocardial infarction in the last 3 months prior to study inclusion or debut of pericarditis;
10. Traumatic chest injury in the last 3 months prior to study inclusion or pericarditis debut;
11. Absence of an informed consent form signed by the patient for participation in the study

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Anonymous male and female patients over 18 years of age suffering from recurrent pericarditis without an established etiology at the time of inclusion in the study (suspected "idiopathic recurrent pericarditis") or diagnosed with "idiopathic recurrent pericarditis"
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-09-30 (Actual); Primary Completion 2028-07-30 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Number of pericarditis recurrences | 6, 12, 18, 24, 30, 36 month
  according to the 2022 nation criteria: intermittent or intermittent (with asymptomatic periods without the use of therapy for more than 6 weeks); continuous-relapsing (discontinuation or reduction in the intensity of anti-inflammatory therapy results in relapse in less than 6 weeks

SECONDARY OUTCOMES:
Number of participants with therapy changes during the past period | 6, 12, 18, 24, 30, 36 month
  Determining therapy changes in patients with recurrent pericarditis at each visit (6, 12, 18, 24, 30, 36 month)
Hospitalization for any reason | 6, 12, 18, 24, 30, 36 month
  To estimate hospitalization for any reason at each visit (6, 12, 18, 24, 30, 36 month) in a cohort of patients with recurrent pericarditis
Hospitalization due to pericarditis | 6, 12, 18, 24, 30, 36 month
  To estimate hospitalization due to pericarditis at each visit (6, 12, 18, 24, 30, 36 month) in a cohort of patients with recurrent pericarditis
Hospitalization for another cardiac cause | 6, 12, 18, 24, 30, 36 month
  To estimate hospitalization for another cardiac cause at each visit (6, 12, 18, 24, 30, 36 month) in a cohort of patients with recurrent pericarditis
Death from any cause | 6, 12, 18, 24, 30, 36 month
  To estimate death from any cause at each visit (6, 12, 18, 24, 30, 36 month) in a cohort of patients with recurrent pericarditis
Death due to cardiac cause | 6, 12, 18, 24, 30, 36 month
  To estimate death due to cardiac cause at each visit (6, 12, 18, 24, 30, 36 month) in a cohort of patients with recurrent pericarditis
Cardiovascular events (STEMI, MI, TIA, etc.) | 6, 12, 18, 24, 30, 36 month
  To assess the development of cardiovascular events in patients with recurrent pericarditis at each visit (6, 12, 18, 24, 30, 36 month)
Development of complications of recurrent pericarditis (constrictive pericarditis, cardiac tamponade, etc.) | 6, 12, 18, 24, 30, 36 month
  To assess the development of complications of recurrent pericarditis in patients with recurrent pericarditis at each visit (6, 12, 18, 24, 30, 36 month)
Quality of life (prospective branch only) | 0, 12, 24, 36 month
  To assess the quality of life of patients with recurrent pericarditis. The quality of life will be assessed using the SF-12 short form, consisting of 12 questions. A low quality of life corresponds to scores of 36-47 points, medium to 24-35 points, and high to 12-23 points.
Pain scale (prospective branch only) | 0, 12, 24, 36 month
  To assess the level of pain (on a pain scale) of patients with recurrent pericarditis. The pain syndrome will be assessed using the Visual Analog Scale, where 10 points indicate unbearable pain and 0 points indicate no pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Eurasian Association of Therapists, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No